CLINICAL TRIAL: NCT00772421
Title: Stimulation of the Anterior Nucleus of the Thalamus for Epilepsy - Recruitment Rhythm (SANTE RR)
Brief Title: Stimulation of the Anterior Nucleus of the Thalamus for Epilepsy - Recruitment Stimulation of the Anterior Nucleus of the Thalamus for Epilepsy - Recruitment Rhythm
Acronym: SANTE RR
Status: Completed | Type: Observational
Sponsor: MedtronicNeuro (Industry)
Responsible Party: Sponsor
Other Study IDs: 1636
Record Dates: First submitted 2008-10-14; First posted 2008-10-15 (Estimated); Last update posted 2012-01-31 (Estimated); Status verified 2012-01

CONDITIONS: Epilepsy
Keywords: Epilepsy; Recruitment rhythm; DBS
MeSH Terms: conditions — Epilepsy

STUDY DESIGN:
Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (2):
- Responder: A subject having at least a 50% reduction in total seizure frequency compared to the SANTE study 3-month Baseline Phase
  Interventions: Device: There was no intervention.
- Non-responder: A subject with a less than 50% reduction in total seizure frequency compared to the SANTE study 3-month Baseline Phase.
  Interventions: Device: There was no intervention.

INTERVENTIONS:
Device: There was no intervention. — There was no intervention. This study was designed as an in-clinic testing protocol to identify recruitment rhythms.

SUMMARY:
The primary objective is to demonstrate that a higher proportion of responders to deep brain stimulation (DBS) in the anterior nucleus (AN) of the thalamus in refractory epilepsy patients in the SANTE study exhibit a recruitment rhythm relative to non-responders.

ELIGIBILITY:
Inclusion Criteria:

* Enrolled in the SANTÉ study, have been implanted with a complete DBS system, and is currently receiving stimulation in the long-term follow-up phase (post Month 13) of the study
* Patient or legal representative is able to understand and provide signed consent for participating in the study
* Willing and available to attend the visit as scheduled and to comply with the study protocol

Exclusion Criteria:

* Patients unable to tolerate stimulation turned OFF during the testing period
* Are pregnant or suspected of being pregnant

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: The study will enroll the number of patients necessary to achieve the required sample size of 18 responders and 18 non-responders at a minimum of six (6) centers participating in the U.S. SANTE study.
Sampling Method: Non-Probability Sample
Enrollment: 29 (Actual)
Dates: Start 2009-01; Primary Completion 2010-05 (Actual); Study Completion 2010-05 (Actual)

PRIMARY OUTCOMES:
To demonstrate that a higher proportion of DBS responders exhibit a RR relative to non-responders, using maximum tolerated voltage settings, at activated electrode contacts used for DBS stimulation in the SANTE study. | Study testing to occur during the long-term follow-up phase of the SANTE trial.

SECONDARY OUTCOMES:
For patients without a RR at their activated DBS electrode contacts used in the SANTE study, demonstrate that activating other electrode contacts generates a RR. | Study testing to occur during the long-term follow-up phase of the SANTE trial.